CLINICAL TRIAL: NCT05325086
Title: Effect on Quality of Life of Information Aimed at Reducing the Impact of a Personality Trait (Openness to Experiences) Identified as a Risk of Non-response to Pulmonary Rehabilitation in Patients With Chronic Respiratory Diseases
Brief Title: Effect on Quality of Life of Adapted Information in Pulmonary Rehabilitation in Chronic Respiratory Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MONTREHAL-1
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Respiratory Disease
Keywords: Pulmonary rehabilitation; Personality traits; Adapted information

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted information arm (Experimental): In parallel with an inpatient PR program, 4 visits will be carried out: V0 : Inclusion / V1 : Randomization / V2 : Follow-up / V3: End-stay.
  At V1:
  * Adapted information to the characteristics of a greater openness to experiences will be delivered to patient.
  * The following questionnaires will be filled : Big Five Inventory BFI-FR, St. George's Respiratory SGRQ, Dyspnea-12, Self-efficacy for managing chronic disease SEMCD-6, Brief Illness Perception B-IPQ, COPD Anxiety Revised CAF-R, Patient Health PHQ-9, Montreal Cognitive Assessment Mini-MoCA
  At V2:
  *Semi-structured individual interviews will be performed. Questions will relate to the information distributed during V1 (adapted information), allowing to assess the understanding and the appropriation of it.
  At V3:
  * The following questionnaires will be filled: SGRQ,Dyspnea-12,SEMCD-6,B-IPQ,CAF-R
  * In addition, some questions will be asked to verify the adherence to information and the potential contamination bias
  Interventions: Other: Adapted information arm
- Neutral information arm (Sham Comparator): In parallel with an inpatient PR program, 4 visits will be carried out: V0 : Inclusion / V1 : Randomization / V2 : Follow-up / V3: End-stay.
  At V1:
  * Neutral information will be delivered to patient.
  * The following questionnaires will be filled : Big Five Inventory BFI-FR, St. George's Respiratory SGRQ, Dyspnea-12, Self-efficacy for managing chronic disease SEMCD-6, Brief Illness Perception B-IPQ, COPD Anxiety Revised CAF-R, Patient Health PHQ-9, Montreal Cognitive Assessment Mini-MoCA
  At V2:
  *Semi-structured individual interviews will be performed. Questions will relate to the information distributed during V1 (neutral information), allowing to assess the understanding and the appropriation of it.
  At V3:
  * The following questionnaires will be filled: SGRQ,Dyspnea-12,SEMCD-6,B-IPQ,CAF-R
  * In addition, some questions will be asked to verify the adherence to information and the potential contamination bias
  Interventions: Other: Neutral information arm

INTERVENTIONS:
Other: Adapted information arm — A adapted booklet will be delivered to patients at the start of the stay. This booklet contains adapted information about the pulmonary rehabilitation targetting the characteristics of the openness to experiences personality traits
  Arms: Adapted information arm
Other: Neutral information arm — A neutral booklet will be delivered to patients at the start of the stay. This booklet contains neutral information about the pulmonary rehabilitation
  Arms: Neutral information arm

SUMMARY:
The purpose of the clinical study is to study the effect of health-related quality of Life of information aimed at reducing the impact of a personality trait (openness to experiences) identified as a risk of non-response to pulmonary rehabilitation in patients with chronic respiratory diseases. This study will determine if a specific information focusing on characteristics of openness to experiences personality trait will lead to better benefits than a general information.

DETAILED DESCRIPTION:
According to the Five Factor Model, personality is made of five dimensions present in varying degrees in individuals and influencing their behavior and life experiences. Several studies showed that some personality traits, according to their level, may positively or negatively influence the quality of life. They can also have an impact on the benefits obtained at the end of one treatment. In the particular context of pulmonary rehabilitation (PR) which is one of the most efficient treatment in respiratory diseases, it has been showed that with a classical support, higher scores for openness to experiences represent a risk factor for non-response in PR on quality of life (i.e. no improvement). Several authors showed that adapted interventions (ex: simple information booklets), based on personality traits, can enhance the effectiveness of the intervention.

Considering that in chronic respiratory diseases, openness to experiences when it is more marked represents a risk of not improving the quality of life following a PR program, the idea of offering information in line with the characteristics of these people (i.e., search for novelties, autonomy, broad and varied interests, etc.) seems relevant and feasible.

The investigators hypothesize that the patients receiving an adapted information aimed at reducing the impact of a personality trait (openness to experiences) will better improve their quality of life in comparison with the patients receiving a neutra information.

The main objective is to assess the impact of life of an adapted information during pulmonary rehabilitation on quality in patients with chronic respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

Admitted for a 4-week inpatient pulmonary rehabilitation program Chronic respiratory disease diagnosis 18 and 80 years old Reading and writing skills Oral consent

Exclusion Criteria:

Inability to participate to exercise training Inability to answer a questionnaire Severe or unstable heart disease, orthopedic, neurologic or psychiatric comorbidities Recent exacerbation (<4 weeks) Pregnant and breastfeeding women Protected adults, pregnant women Participation in another study, with the exception of observational studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Differential of health-related quality of life from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of health-related quality of life score on St. George's Respiratory Questionnaire (SGRQ) (Jones et al., 1991) from baseline to PR end-stay within and between groups
  The SGRQ contains 50 questions and evaluates 3 dimensions : symptoms component, activities that cause or are limited by breathlessness and impact component

SECONDARY OUTCOMES:
Differential of dyspnea from from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of dyspnea score on DYSPNEA-12 questionnaire (Yorke et al 2010) within and between groups.
  The Dyspnea-12 contains 12items and evaluate the physical and affective dimensions of dyspnea.
Differential of exercise tolerance from from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of exercise tolerance on the 6-minute walking test within and between groups.
Differential of self-efficacy from from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of self-efficacy score on Self-efficacy for managing chronic disease SEMCD-6 questionnaire (Ritter & Lorig, 2014) within and between groups. This questionnaire contains 6 items.
Differential of disease-related thinking from from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of disease-related thinking score on Brief Illness Perception Questionnaire B-IPQ (Broadbent et al., 2006) within and between groups.
  This questionnaire contains 8 items.
Differential of disease-related fears from from baseline to PR end-stay | Changes from baseline (T0) to at the end of the 4-weeks PR (T1)
  Assessing differential of disease-related fears score on COPD Anxiety Questionnaire Revised CAF-R (Keil et al., 2014) within and between groups.
  This questionnaire contains 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin EICHENAUER, Principal Investigator — Korian; Nelly HERAUD, Study Director — Korian; Brice CANADA, Study Director — Université de Lyon
Locations (2):
- France (2):
  - Clinique du Souffle le Pontet, Hauteville-Lompnes
  - Clinique du Souffle Les Clarines, Riom-ès-Montagnes

IPD SHARING:
Plan to Share IPD: No